CLINICAL TRIAL: NCT00042224
Title: ECT in Clozapine Refractory Schizophrenia
Brief Title: Electroconvulsive Therapy in Clozapine Refractory Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, George Petrides, Associate Professor of Psychiatry, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH060390 (NIH); R01MH060390 (NIH); DSIR AT-SO (Other: NorthShore LIJ Health System)
Record Dates: First submitted 2002-07-24; First posted 2002-07-26 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia
Keywords: Electroconvulsive Therapy
MeSH Terms: conditions — Schizophrenia | interventions — Electroconvulsive Therapy; Clozapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 ECT plus clozapine (Experimental): Electroconvulsive therapy ECT plus clozapine for 8 weeks
  Interventions: Procedure: Electroconvulsive Therapy (ECT); Drug: Clozapine
- 2 Clozapine (Active Comparator): Clozapine for 8 weeks
  Interventions: Drug: Clozapine

INTERVENTIONS:
Procedure: Electroconvulsive Therapy (ECT) — ECT will be used to augment clozapine in schizophrenic patients who continue to have psychotic symptoms despite optimal treatment with clozapine.
  Arms: 1 ECT plus clozapine
Drug: Clozapine — Patients with psychotic symptoms will receive clozapine
  Other Names: Clozaril

SUMMARY:
This study will evaluate electroconvulsive therapy (ECT) in patients who have not responded adequately to clozapine.

DETAILED DESCRIPTION:
ECT augmentation of clozapine will be compared to clozapine monotherapy in schizophrenic patients who continue to have psychotic symptoms despite optimal treatment with clozapine.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of schizophrenia according to DSM-IV criteria
* Duration of illness 2 years or greater
* Resistance to at least 2 antipsychotics
* Clozapine resistance
* Capacity to give informed consent
* For women of childbearing capacity, a negative pregnancy test and patient agreement to use a medically accepted form of contraception
* Brief Psychiatric Rating Scale score of at least a 4 on one of the four psychotic items on the psychotic sub-scale or a score of 12 on these 4 items combined.
* Clinical Global Impressions (CGI) - severity rating of at least moderate (score of 4)
* Receiving at least two 400 mg doses of chlorpromazine equivalents for at least 4 weeks (may include newer antipsychotics)
* Having substantial psychotic symptoms despite at least 12 weeks of treatment (at least 8 weeks at a consistent dose)

Exclusion criteria

* schizoaffective disorder; bipolar disorder;
* current affective episode;
* Electroconvulsive Therapy (ECT) within the past 6 months
* history of epilepsy; severe neurological or systemic disorder that could significantly affect cognition, behavior, or mental status (other than tardive dyskinesia or neuroleptic-induced parkinsonism); psychoactive substance dependence (other than nicotine or caffeine) within 1 month prior to entering the study
* a score of less than 18 on the 24-item Hamilton Depression Rating Scale (HAM-D)
* clinical determination that mood stabilizers were necessary and therefore could not be discontinued.
* pregnancy.
* affective disorders and prominent depressive symptoms because ECT is well known to be effective in those situations, and we wanted to avoid contamination of our results by improvement solely driven by the treatment of the affective symptoms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2000-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Petrides, MD, Principal Investigator — New Jersey Medical School
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited from the inpatient units of the Zucker Hillside Hospital at Glen Oaks, N.Y., and the Pilgrim State Psychiatric Center in Long Island, N.Y.
Pre-assignment Details: In an 8-week random-assignment study incorporating nonblinded treatment and blinded assessments, patients with antipsychotic and clozapine-resistant schizophrenia were assigned to two treatment groups.
Groups:
- 1 Electroconvulsive Therapy With Medication: Electroconvulsive Therapy (ECT): ECT will be used to augment clozapine in schizophrenic patients who continue to have psychotic symptoms despite optimal treatment with clozapine.
  Clozapine: Patients with psychotic symptoms will receive clozapine
- 2 Medication Monotherapy: Clozapine: Patients with psychotic symptoms will receive clozapine
Period: Overall Study
Arm/Group | 1 Electroconvulsive Therapy With Medication | 2 Medication Monotherapy
Started | 20 | 19
Completed | 17 | 16
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Electroconvulsive Therapy With Medication: Procedure/Surgery: Electroconvulsive Therapy (ECT) ECT will be used to augment clozapine in schizophrenic patients who continue to have psychotic symptoms despite optimal treatment with clozapine.
  Drug: Clozapine Patients with psychotic symptoms will receive clozapine
  Other Names:
  • Clozaril
- Medication Monotherapy: Drug: Clozapine Patients with psychotic symptoms will receive clozapine
  Other Names:
  • Clozaril
- Total: Total of all reporting groups
Arm/Group | Electroconvulsive Therapy With Medication | Medication Monotherapy | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.70 (2.27) | 42.78 (1.82) | 39.24 (2.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 18
  Male | 15 | 6 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Response Rates in the ECT Plus Clozapine Group vs the Pharmacotherapy Group.
Description: Response is defined as 40% reduction of symptoms in the psychotic symptom sub-scale (hallucinatory behavior, suspiciousness, conceptual disorganization, and unusual thought of content) of the Brief Psychiatric Rating Scale (BPRS) at the end of the 8-week study. BPRS assesses psychotic symptoms on a 18-item scale. The severity of each item is rated on a continuous scale from 1-7, with 1 being the least severe and 7 being most severe. Participants included in the study, at baseline had at least a moderate score of 4 on one of the four psychotic symptom sub-scale or a score of 12 on all four of these items combined (ranges 4 -28, with higher scores indicative of greater severity). A reduction of symptoms would be a sub-scale score which is 40% less than participants baseline score. If a participant enters the study with a sub-scale score of 15, to be considered a responder (at least a 40% reduction in symptoms score) his/her score must decrease by at least 6 points and be 9 or less.
Time Frame: 8 Weeks
Population: inpatient units of the Zucker Hillside Hospital at Glen Oaks, N.Y., and the Pilgrim State Psychiatric Center in Long Island, N.Y.
Measure: Number; unit: Percentage of responders
Arm/Group | Electroconvulsive Therapy With Medication | Medication Monotherapy
Number analyzed (Participants) | 20 | 19
Percentage of responders | 50 | 0

ADVERSE EVENTS:
Arm/Group | Electroconvulsive Therapy With Medication | Medication Monotherapy
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes